CLINICAL TRIAL: NCT04698668
Title: Fusion Radiology in Interventional Endoscopy (FRIEnd) Approach for Pancreatic Fluid Collections
Brief Title: Evaluation of the Outcomes and Performances of the Application of Augmented Reality in Operative Digestive Endoscopy
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: GASTRO.04.2020
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2021-02

CONDITIONS: Pseudocyst; Walled Off Cavity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1: Patients with pancreatic fluid collection treated with traditional EUS-drainage
- 2: Patients with pancreatic fluid collection treated with fusion imaging
  Interventions: Device: fusion imaging

INTERVENTIONS:
Device: fusion imaging — To drain a pancreatic fluid collection through the assitance of the CT-scan image that is superimposed on the radiological field
  Groups: 2

SUMMARY:
Virtual reality obtained by the fusion of images can be applied to several fields of medicine leading to the so called "augmented reality". Since 2017 investigators have been using a new digital angiographic system (Discovery IGS 40, General Electrics), where fluoroscopy can be fused with pre-procedural CT o MRI. Specifically the present study aimed at verifying the advantages that fusion imaging could bring in EUS-guided drainage of post-pancreatitis fluid collection (PFC), i.e. pseudocysts or WON, in terms of more appropriate visualization, drainage approach and time needed for resolution.

DETAILED DESCRIPTION:
17 drainages performed with traditional radiology (group 1) were retrospectively compared with 14 ones achieved with the fusion approach (group 2). The two population were homogenous for age, sex, pancreatitis etiology and indication for drainage whereas PFCs of group 2 were larger (663 cm3 vs 437 cm3), more frequently WON than pseudocysts and were treated more precociously. As for procedure, in the group 2, thanks to fusion imaging, endoscopists didn't need ever contrast media - that was pivotal with traditional radiology - to adequately define lesion morphology. LAMS (Axios) stents were placed mainly in group 2, while in group 1 other types of stent were used.

ELIGIBILITY:
Inclusion Criteria:

* patients with post-pancreatitis PCF endoscopically drained

Exclusion Criteria:

* refuse to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient affected by moderate-severe pancreatits whio develops a PFC (WON or pseudocysts) that requires an endoscopic drainage
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
clinical and radiological resolution of the PFC | 12 months
  complete emtying of the PFC tighter with resolution of patients' symptomps
time of radiological resolution | 12 months
  time taken for the complete emtying of the PFC

CONTACTS AND LOCATIONS:
Overall Officials: Romano Sassatelli, Study Director — IRCCS-AUSL Reggio Emilia
Locations (1):
- IRCCS-AUSL Reggio Emilia, Reggio Emilia, RE, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Arvanitakis M, Dumonceau JM, Albert J, Badaoui A, Bali MA, Barthet M, Besselink M, Deviere J, Oliveira Ferreira A, Gyokeres T, Hritz I, Hucl T, Milashka M, Papanikolaou IS, Poley JW, Seewald S, Vanbiervliet G, van Lienden K, van Santvoort H, Voermans R, Delhaye M, van Hooft J. Endoscopic management of acute necrotizing pancreatitis: European Society of Gastrointestinal Endoscopy (ESGE) evidence-based multidisciplinary guidelines. Endoscopy. 2018 May;50(5):524-546. doi: 10.1055/a-0588-5365. Epub 2018 Apr 9. PMID 29631305
- [Background] Rajagopal M, Venkatesan AM. Image fusion and navigation platforms for percutaneous image-guided interventions. Abdom Radiol (NY). 2016 Apr;41(4):620-8. doi: 10.1007/s00261-016-0645-7. PMID 26826086
- [Background] Zhang H, Chen GY, Xiao L, Ma X, Shi L, Wang T, Yan HT, Zou H, Chen Q, Tang LJ, Liu WH. Ultrasonic/CT image fusion guidance facilitating percutaneous catheter drainage in treatment of acute pancreatitis complicated with infected walled-off necrosis. Pancreatology. 2018 Sep;18(6):635-641. doi: 10.1016/j.pan.2018.06.004. Epub 2018 Jun 18. PMID 29954676
- [Background] ASGE Standards of Practice Committee; Early DS, Acosta RD, Chandrasekhara V, Chathadi KV, Decker GA, Evans JA, Fanelli RD, Fisher DA, Fonkalsrud L, Hwang JH, Jue TL, Khashab MA, Lightdale JR, Muthusamy VR, Pasha SF, Saltzman JR, Sharaf RN, Shergill AK, Cash BD. Adverse events associated with EUS and EUS with FNA. Gastrointest Endosc. 2013 Jun;77(6):839-43. doi: 10.1016/j.gie.2013.02.018. No abstract available. PMID 23684089